CLINICAL TRIAL: NCT06452888
Title: Improvement of Medical Quality and Outcomes Through Intelligent Management and Decision System of Cerebrovascular Diseases Based on Hospital Information System - A Multicenter, Open-label, Cluster-Randomized Controlled Study
Brief Title: Improvement of Medical Quality and Outcomes Through Intelligent Management and Decision System of Cerebrovascular Diseases Based on Hospital Information System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zi-Xiao Li, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022YFC2504902
Record Dates: First submitted 2024-05-21; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cerebrovascular Disease
Keywords: Ischemic Stroke; Medical Quality; Clinical Complication; Clinical decision Support System; Electronic Health Record; Artificial Intelligence
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (Sham Comparator): The control group indicated that the physicians will not be provided with the information of multifaceted improvement tools including evidence-based clinical pathway, standard operating procedures (SOP) of performance indicators a quality coordinator, and monitoring and feedback system of performance measures. They just provide patients with routine care.
  Interventions: Behavioral: no intervention
- Intervention Group (Experimental): Patients in the intervention group will receive the organizational management based clinical decision support system, including evidence-based clinical pathway, standard operating procedures (SOP) of performance indicators, a quality coordinator, and monitoring and feedback system of performance measures.
  Interventions: Behavioral: Clinical decision support system.

INTERVENTIONS:
Behavioral: Clinical decision support system. — The clinical decision support system includes evidence-based clinical pathway, standard operating procedures (SOP) of performance indicators, a quality coordinator, and monitoring and feedback system of performance measures. Patients in the intervention group will receive the organizational management based on the guidelines and conduct intervention management for patients with actue ischemic stroke. The clinical decision system will classify the patients into risk factors, automatically generate treatment measures according to the guidelines, in order to standardize the treatment of physicians. Such as the management of complications after stroke, the treatment of antiplatelet, anticoagulation, antihypertensive and hypoglycemic.
  Arms: Intervention Group
Behavioral: no intervention — No intervention indicated that the physicians among control hospital provide routine
  Arms: No intervention

SUMMARY:
This study applied a cerebrovascular disease organizational management and decision system based on hospital information system, aiming to verify the effect of intervention and management after stroke on improving the functional outcomes of acute ischemic cerebrovascular disease through a cluster randomized controlled study.

DETAILED DESCRIPTION:
Stroke is a major cerebrovascular disease that causing high morbidity, disability and mortality. Management of the acute phase of stroke is critical to functional outcomes. Our study aims to verify an intervention method based on hospital information management decision system for the prevention and management of post-stroke treatment in acute stroke patients and improve long-term functional prognosis.

This study was a multicenter, open-label, parallel, cohort randomized controlled study, recruiting acute ischemic stroke patients with a post-onset National Institutes of Health Stroke Scale (NIHSS) score of ≥ 2 (limb score ≥1) within 7 days from onset of symptoms. This study will recruit a total of 3540 patients in 30 secondary hospitals. Patients in the intervention group will receive the organizational management based clinical decision support system recommended by the guidelines and conduct intervention management for patients with acute ischemic stroke. All patients in control group were treated with conventional diagnosis and treatment. The primary endpoint event was unfavorable functional outcome 3 months after onset. Secondary outcomes were in-hospital complications (including pneumonia, deep vein thrombosis), unfavorable functional outcomes at 6 and 12 months of onset (Modified Rankin Score (mRS) Score 2-5), recurrent stroke at 3, 6, and 12 months, new vascular events (including ischemic stroke, hemorrhagic stroke, myocardial infarction or vascular death) and all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* Diagnosed with ischemic stroke confirmed by magnetic resonance imaging (MRI) or brain computed tomography (CT).
* Within 7 days from onset of symptoms.
* With a NIHSS score of ≥2 at admission (limb score ≥1).
* With a prestroke mRS score of 0-1.
* Admission from the emergency department or outpatient service.
* Voluntary informed consent.

Exclusion Criteria:

* Diagnosis of other cerebrovascular diseases (cerebral hemorrhage, subarachnoid hemorrhage, cerebral venous sinus thrombosis, etc.).
* Diagnosis of non-cerebrovascular disease (central nervous system infection, epilepsy, metabolic encephalopathy, etc.).
* Ischemic stroke with negative diffusion weighted imaging (DWI).
* Being tested for interventions such as drugs or instruments.
* Pregnancy or 6 weeks postpartum.
* With a life expectancy of less than 3 months or who were unable to complete the study follow-up for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3540 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of unfavorable functional outcome | Participants will be followed at 3 months after enrollment.
  Unfavorable functional outcome is defined as the modified Rankin Scale (mRS) Score 2-5. mRS is an efficient, reliable and simple scale to assess the recovery of neurological function and disability after stroke. The high score indicates the poor neurological recovery. The minimum score (0) means no symptoms at all. The maximum (6) means death.

SECONDARY OUTCOMES:
The incidence of in-hospital complications | Participants will be followed at 3, 6 and 12 months after enrollment.
  In-hospital complications (including pneumonia, deep vein thrombosis, gastrointestinal bleeding, and urinary tract infection).
The incidence of unfavorable functional outcome | Participants will be followed at 6 and 12 months after enrollment.
  Unfavorable functional outcome is defined as the modified Rankin Scale (mRS) Score 2-5. mRS is an efficient, reliable and simple scale to assess the recovery of neurological function and disability after stroke. The high score indicates the poor neurological recovery. The minimum score (0) means no symptoms at all. The maximum (6) means death.
The incidence of new vascular events | Participants will be followed at 3, 6 and 12 months after enrollment.
  Including ischemic stroke, hemorrhagic stroke, myocardial infarction or vascular death.
The incidence of recurrent ischemic stroke | Participants will be followed at 3, 6 and 12 months after enrollment.
  Stroke recurrence is defined as a new focal neurological impairment that was confirmed by neuroimaging, including both ischemic stroke and hemorrhagic stroke.
The incidence of all-cause death | Participants will be followed at 3, 6 and 12 months after enrollment.
  An all-cause death is defined as a death from any cause.
The incidence of moderate or severe bleeding events | Participants will be followed at 3, 6 and 12 months after enrollment.
  Defined by the Global Utilisation of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO).
The incidence of all bleeding events | Participants will be followed at 3, 6 and 12 months after enrollment.
  Including moderate or severe bleeding events, gastrointestinal bleeding, mucocutaneous hemorrhage, respiratory system bleeding and other.

OTHER OUTCOMES:
The incidence of average length of stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  The average length of stay of all patients enrolled in the subcenter.
The incidence of average total hospital expenses | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  The average total hospital expenses of all patients enrolled in the subcenter.